CLINICAL TRIAL: NCT00203866
Title: A Randomized Pilot Phase II Trial of Adjuvant Immunization With G250 Peptide andThree Different Dose Levels of IL-2 Following Surgical Resection of Locally Advanced or Metastatic Renal Cell Carcinoma
Brief Title: Trial of G250 Peptide and IL-2 Following Surgical Resection of Locally Advanced/Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study completed
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12403B
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: G250 peptide
Drug: IL-2

SUMMARY:
The purpose of this study is to determine whether the experimental vaccine G250 with or without IL-2 can produce an immune response in patients with renal cell carcinoma who have had all their cancer removed by surgery.

DETAILED DESCRIPTION:
Renal cell carcinoma is a chemotherapy and radiotherapy resistant neoplasm that has a poor prognosis. Immunotherapy with the biologic agent IL-2 consistently produces a response rate of 10-15 %. Currently, for patients with locally advanced disease or patients with solitary metastases, the only treatment modality with a curative potential is surgical resection. There is presently no approved agent for use as adjuvant therapy after surgical resection to decrease the risk of recurrence. Peptide-based vaccine approaches offer an attractive treatment option.

The high prevalence of G250 in RCC, the definition of an HLA-A2-restricted epitope (the most common HLA type), and its immunogenicity makes it the most attractive candidate for peptide-based vaccine approaches in RCC therapy. The promising preclinical and clinical evidence provides the rationale for the use of IL-2 to potentiate the antitumor effects of cancer vaccines.

There is presently no conclusive data on the best dose of IL-2 to use as an adjuvant to cancer vaccines. One paradoxical finding in preclinical and clinical trials is that despite the enhancement in the antitumor effects of cancer vaccines, the number of antigen-specific CTL is not increased when IL-2 is given with a cancer vaccine 35]. In contrast, patients treated with peptide vaccines (without IL-2) in some melanoma trials had evidence of high levels of antigen-specific CTL, with no tumor regression observed 36]. Some possible explanations include capillary leak from high dose IL-2 resulting in CTL leaving the circulation and the possibility that high dose IL-2 decreases efficient T-cell priming. A more recent explanation has been proposed through advances in the mechanism of 1-cell activation. As their level of activation increases, T-cells become more susceptible to apoptosis. This phenomenon is known as activation-induced cell death (AICD) IL-2 may then have a role in the amplification and downregulation of the immune response. High dose IL-2 may help in augmenting the increase in the activation of CTL, but this may lead to increase their susceptibility to AJCD. The evidence in animal models that low doses of IL-2 were sufficient in increasing the potency of DC-based immunizations provides the rational for our study.

In our current study, the lowest dose of IL-2 (1 x 106 IU) is similar to the doses used by Yee et al. in their adoptive I cell therapy. This dose has been shown to expand and maintain CTLs in both preclinical and clinical models. The highest dose (11 x 106 IU) was chosen based on the expected toxicities from higher doses of IL-2 and our experience with this dose as a single agent in RCC.

Our hypothesis is that immunization with G250/Montanide/GM-CSF plus IL-2 can lead to an expansion of G250-specific CTL and result in killing of 0250 expressing micrometastatic RCC. We propose a dose finding study of escalating low doses of IL 2 (subcutaneous), since no prior study has specifically evaluated the use of low dose IL-2 as a cytokine adjuvant and attempted to establish a correlation between dose and immunolgic response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must express HLA-A2
* Patients must have histologically or cytologically proven renal cell carcinoma that expresses G250 by IHC
* Patients must have completely resected disease without any evidence of residual local or metastatic disease
* Patients with resected locally advanced disease
* Patients with metastatic disease(including synchronous metastatic site)
* Patients with solitary metachronous metastatic disease
* Age >/=18 years
* ECOG performance status 0-1
* Patients must have normal organ and marrow function
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, or an experimental (investigational) agent prior to starting treatment. Prior biologic therapy (IL-2 or interferon) is allowed only if it precedes a curative surgical therapy.
* Patients may not have received a previous G250 vaccine.
* Patients with residual metastatic disease following surgical resection are excluded from this clinical trial.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to G250, Montanide ISA-5 1, OM-CSF, or IL-2.
* Patients must not have autoimmune disorders (SLE, Rheumatoid Arthritis), conditions of immunosuppression (such as HIV), or treatment with immunosuppressive drugs (including oral steroids, continuous use of topical steroids, steroid inhalers). Replacement doses of steroids for patients with adrenal insufficiency are allowed.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active GI bleeding, inflammatory bowel disease or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast-feeding women
* HIV-positive patients
* Patients with a currently active second malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix are not to be registered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To determine whether immunization with G250 peptide/Montanide/GM-CSF plus IL-2 elicits a specific CTL response as assessed by ELISPOT.

SECONDARY OUTCOMES:
To explore differences in G250-specific CTL response as a function of IL-2 dose.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States